CLINICAL TRIAL: NCT06137612
Title: Spinal Cord Gray Matter Imaging - a Novel Biomarker for Spinal Muscular Atrophy - a Pilot Study
Brief Title: Spinal Cord Gray Matter Imaging in Spinal Muscular Atrophy
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: SMA_SC_Imaging_1
Record Dates: First submitted 2023-11-08; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Spinal Muscular Atrophy Type III; Spinal Muscular Atrophy Type II
MeSH Terms: conditions — Spinal Muscular Atrophies of Childhood

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with SMA: Patients with SMA type II and III
  Interventions: Diagnostic Test: MRI
- Healthy controls: Age- and sex-matched HC
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — axial 2D rAMIRA (radially sampled averaged magnetization inversion recovery acquisitions) imaging at selected levels of cervical and thoracic spinal cord at the intervertebral disc levels perpendicular to the spinal cord.

SUMMARY:
This study aims to measure the spinal cord gray matter in patients with spinal muscular atrophy (SMA) type II and III in comparison with age- and sex-matched healthy controls (HC) using rAMIRA (radially sampled averaged magnetization inversion recovery acquisitions) imaging, a novel MRI (Magnetic Resonance Imaging) method. Patient and HC undergo MRI examinations, clinical/neurological (handheld dynamometry) and electrophysiological investigations (MUNIX, Motor Unit Number Index). Serum markers of neuro-axonal and astrocytic injury are also assessed.

DETAILED DESCRIPTION:
Patients with the diagnosis of 5q-SMA (spinal muscular atrophy) types II or III (confirmed by genetic testing) will be recruited. Healthy age and sex-matched controls will also be investigated.

Patients will be neurologically investigated at the Neurology Policlinic, University Hospital Basel, including standard muscle force measurements on the British Medical Council (BMC) grade, and quantitative muscle force tests by hand held dynamometer of selected muscles.

All patients will also complete the SMA functional rating scale (SMA-FRS). Age and sex matched healthy controls will also undergo a standardized neurological examination to ensure that no other neurological condition is present that could potentially interfere with the test results.

All participants will be scanned on the same 3 Tesla MR-Scanner (Magnetom PRISMA, Siemens Healthineers) at the University Hospital Basel. The protocol includes axial 2D rAMIRA imaging at selected levels of cervical and thoracic spinal cord at the intervertebral disc levels perpendicular to the spinal cord, and diffusion tensor imaging (DTI) at selected positions, a standard diagnostic high-resolution T2w sequence of the spinal cord and a high-resolution T1w structural imaging of the brain for cortical/subcortical volumetry.

Serum biomarkers will also be evaluated including serum neurofilament light chain (NfL) levels .

MUNIX is an electrophysiological method that is used in clinical routine in many neuromuscular centers to quantitate the number of functioning motor units. Patients and controls will undergo MUNIX testing .

Patients will be examined by a professional physiotherapist to assess the Motor Function Measure (MFM), Revised Hammersmith Scale for SMA, Revised Upper Limb Module, time to rise from the floor, and 6 minutes walk test.

ELIGIBILITY:
Inclusion Criteria (patients)

1. 11 years or older
2. Informed consent by the participants or, in children below the age of legal consent, by a legally authorized representative
3. genetically confirmed diagnosis of 5q-SMA (Types II or III)

Exclusion Criteria (patients):

1. active other neurological or neuromuscular condition explaining the symptoms or a significant part of it
2. other neurological or neuromuscular conditions interfering with the examinations
3. other severe chronic disease
4. pregnancy
5. general contraindications against MRI scanning (e.g. pacemakers)
6. not able to understand the patient information due to language barriers
7. In the event of a participant incapable of judgment, symptoms showing that the participant is unwilling to participate in the study will result in the participant being excluded from participation

Inclusion Criteria (healthy volunteers)

1. participants will be selected to be age-and sex-matched to the patients
2. 11 years or older
3. Informed consent by the participants or, in children below the age of legal consent, by a legally authorized representative

Exclusion Criteria (healthy volunteers):

1. active neurological or neuromuscular condition
2. other neurological or neuromuscular conditions interfering with the examinations
3. other severe chronic disease
4. pregnancy
5. general contraindications against MRI scanning (e.g. pacemakers)
6. not able to understand the patient information due to language barriers
7. In the event of a participant incapable of judgment, symptoms showing that the participant is unwilling to participate in the study will result in the participant being excluded from participation

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with the diagnosis of 5q-SMA II or III (confirmed by genetic testing) will be recruited. Healthy age and sex-matched controls will also be investigated.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2020-08-17 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Spinal cord gray matter atrophy | baseline
  Difference in spinal cord gray matter (GM) cross-sectional area in mm2 between SMA patients and age and sex matched HC subjects

SECONDARY OUTCOMES:
Associations | baseline
  Cross-sectional associations between spinal cord GM areas (in mm2) and segmental quantitative muscle force (in Newton) in SMA patients
Associations | baseline
  Cross-sectional associations between spinal cord GM areas (in mm2) and SMA-FRS-R Score in SMA patients
Associations | baseline
  Cross-sectional associations between spinal cord GM areas (in mm2) and RULM Score in SMA patients
Associations | baseline
  Cross-sectional associations between spinal cord GM areas (in mm2) and HFSME Score in SMA patients
Associations | baseline
  Cross-sectional associations between spinal cord GM areas (in mm2) and MFM Score in SMA patients
Associations | baseline
  Cross-sectional associations between spinal cord GM areas (in mm2) and serum NfL(pg/ml)
Associations | baseline
  Cross-sectional associations between spinal cord GM areas (in mm2) and MUNIX (Index)
Associations | baseline
  Cross-sectional associations between spinal cord GM areas (in mm2) and 6MWT
Associations | baseline
  Cross-sectional associations between spinal cord GM areas (in mm2) and time to rise from the floor

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided